CLINICAL TRIAL: NCT03591107
Title: Trauma-informed Collaborative Care for Low-income African Americans With Posttraumatic Stress Disorder (PTSD)
Brief Title: Trauma-informed Collaborative Care for Low-income African Americans With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Collaborators: Louisiana Public Health Institute (Other)
Responsible Party: Principal Investigator, Lisa Meredith, Senior Behavioral Scientist, RAND
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34MH111860 (NIH)
Record Dates: First submitted 2018-07-06; First posted 2018-07-18 (Actual); Results first posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Recruitment Coordinators/Data Collectors will only recruit at one of the two sites. The baseline assessment will be conducted prior to random assignment. After the assessment, they will be aware of study assignment which is necessary for connecting patients assigned to the PCM arm to connect patients to the Care Manager. However, they will only conduct 6-month assessments with patients from the "other" site and therefore will not be aware of the assignments for those patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTSD Care Management (PCM) (Experimental): In addition to the education and feedback components for both conditions the PCM intervention provides access to a trained Care Manager (CM) who will engage the patient into care, monitor progress over 6 months, coordinate care with primary care and behavioral healthcare providers and social services, and receive monthly supervision by the study psychiatrist.
  Interventions: Other: PTSD Care Management (PCM)
- Minimally Enhanced Usual Care (MEU) (Active Comparator): The MEU condition will consist of only clinician education, patient education (Information Sheet) and feedback about having a probably diagnosis of PTSD to both the clinician and patient.
  Interventions: Other: Minimally Enhanced Usual Care (MEU)

INTERVENTIONS:
Other: PTSD Care Management (PCM) — Collaborative care for PTSD facilitated by a trained CM who will engage the patient into care, monitor progress over 6 months, coordinate care with primary care and behavioral healthcare providers and social services, and receive monthly supervision by the study psychiatrist in addition to education and feedback
  Arms: PTSD Care Management (PCM)
Other: Minimally Enhanced Usual Care (MEU) — Education and feedback alone
  Arms: Minimally Enhanced Usual Care (MEU)

SUMMARY:
The purpose of this study is to optimize, culturally adapt, implement, and pilot test a trauma-informed collaborative care intervention for low-income African Americans who receive care in Federally Qualified Health Centers (FQHCs) in New Orleans, Louisiana. We will randomize 40 patients to either a Posttraumatic Stress Disorder (PTSD) collaborative care intervention or to an enhanced usual care control and will evaluate the effectiveness of the intervention (including whether outcome expectancy, coping efficacy, and trust mediate the impact of the intervention) as well as its feasibility, tolerability, and acceptability.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is prevalent in the general population, especially among low-income African Americans. Within primary care settings, PTSD may affect as many as one in four patients. PTSD is among the most difficult and costly psychiatric disorders to treat because it is necessary to go beyond traditional medical care to also address the trauma in patients' lives that interferes with treatment and potentially attenuates treatment benefits. African Americans are also less likely to receive care for mental health problems. Several social psychological barriers (e,g., mistrust in healthcare providers, skepticism about treatment efficacy, negative beliefs in one's ability to cope with PTSD), and logistical barriers (e.g., limited access to care, lack of transportation and childcare, lack of financial resources) impede engagement into care. Thus, a trauma-informed approach to care that emphasizes the promotion of trust, safety, self-efficacy, peer support, cultural competency, collaboration, and coordinates with social services in the community to address logistical barriers is required to treat PTSD in low-income African Americans.

Growing evidence suggests that collaborative care for PTSD in primary care is effective. In two studies (Telemedicine-Based Collaborative Care for PTSD (TOP) and Stepped Enhancement of PTSD Services Using Primary CARE (STEPS-UP)) collaborative care significantly improved outcomes relative to usual care and attributed success in large part to the high levels of patient engagement (100%) associated with strategies to connect patients to care including behavioral activation, problem solving, and motivational interviewing. Three trials showed overall improvements but no relative advantage for collaborative care over usual care. The Coordinated Anxiety Learning and Management (CALM) study of anxiety disorders among civilians showed a trend favoring collaborative care (the effect in the PTSD subgroup was not statistically significant due to the insufficient sample size) but engagement was high (95%). Another trial for veterans Re-Engineering Systems for the Primary Care Treatment of PTSD (RESPECT-PTSD) found no difference between arms. Our recently completed Violence and Stress Assessment (ViStA) trial for low-income patients in Federally Qualified Health Centers (FQHCs) also found no differential effect. In both ViStA and RESPECT-PTSD, patient engagement was low - only 73% and 62% of patients initiated treatment, respectively. However, in both studies, use of mental health services was significantly higher among the patients who engaged in collaborative care suggesting that adding strategies to boost engagement would increase its effectiveness. Also in ViStA, prior to the intervention, there were significant disparities in care for the African Americans in our sample with rates of minimally adequate care of only 21% compared to Whites (33%). This suggests that a trauma-informed approach that addresses social psychological and logistical barriers may better engage patients, enhance collaborative care, and ultimately, improve outcomes.

The Institute of Medicine has prioritized effective delivery approaches that engage individuals with PTSD. We propose to optimize, culturally adapt, and pilot test a collaborative care intervention that uses a trauma-informed approach to identify specific target mechanisms to improve treatment engagement, and reduce PTSD diagnosis and symptoms in primary care settings that serve low-income African Americans. Specifically, we will test the effectiveness of collaborative care, optimized based on lessons from previous studies, adapted to be culturally relevant for this population, and will directly address target mechanisms (outcome expectancy, coping efficacy, and trust). All components of collaborative care will be delivered by African American care managers (CMs) with the guidance of a local, African American community workgroup. We will compare this PTSD collaborative care with a CM (PCM) approach to minimally enhanced usual care (MEU). We submit this R34 application in response to RFA-MH-16-410, which elicits pilot effectiveness trials for treatment, preventive and services intervention. This proposal is an excellent fit for this funding opportunity because our intervention has potential to substantially impact practice and public health by improving mental health outcomes among African Americans with PTSD in New Orleans FQHCs using an empirically grounded approach. Our three Specific Aims are to:

Aim 1: Optimize, culturally adapt, and implement an evidence-based trauma-informed model of PTSD collaborative care (PCM) compared with MEU for underserved African Americans. We will recruit patients at two FQHCs in New Orleans, LA to assess the feasibility, tolerability, and acceptability of PCM.

Aim 2: Conduct a pilot randomized trial of the optimized/adapted PCM intervention compared with MEU in two FQHCs with 40 African American patients to evaluate its impact on social psychological target mechanisms - outcome expectancy, coping efficacy, and trust in facilitating treatment engagement.

Aim 3: Evaluate the effectiveness of the PCM intervention (compared with MEU) on outcomes - PTSD diagnosis and symptoms (primary outcomes) and use of mental health care and non-medical community services and resources (secondary outcomes) either directly or indirectly as mediated by the target mechanisms before and one year after the start of the intervention.

Preliminary data from this pilot effectiveness trial will pave the way for a larger-scale intervention.

ELIGIBILITY:
Inclusion Criteria:

* Have a scheduled or walk-in appointment with a primary care provider at the clinic
* Age 18 or over
* Self-identify as African American
* Consider clinic their usual source of care
* No physical or cognitive disabilities that would preclude completing assessments

Exclusion Criteria:

* Does not screen positive for probable PTSD on the PCL-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-10-12 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa S Meredith, PhD, Principal Investigator — RAND
Locations (1):
- EXCELth Family Health and Dental 70127New Orleans East, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We completed patient recruitment across 70 days over the course of nine months from October 12, 2018, to July 2, 2019. Patients were approached in the primary care waiting area and if they met inclusion criteria they were asked to complete a brief PTSD symptom checklist, followed by a longer PTSD assessment. If patients met criteria for a provisional diagnosis of PTSD, they were invited to enroll in the study and asked for informed consent (n= 42) adult patients.
Period: Overall Study
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
Started | 21 | 21
Completed | 20 | 16
Not Completed | 1 | 5
Not completed — Same patient in both arms | 1 | 1
Not completed — Sought care at other clinics | 0 | 2
Not completed — Discharged from clinic | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU) | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 21 | 40
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 3 | 5 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 19 | 21 | 40
Education [Count of Participants; unit: Participants]
  < High school | 2 | 10 | 12
  High school graduate/GED | 8 | 9 | 17
  College degree or graduate | 9 | 2 | 11
Marital status [Count of Participants; unit: Participants]
  Single | 13 | 10 | 23
  Married or unmarried couple | 1 | 3 | 4
  Separated/divorced/widowed | 5 | 8 | 13
Type of medical insurance [Count of Participants; unit: Participants]
  Medicaid | 15 | 18 | 33
  Medicare | 2 | 1 | 3
  Employer/private | 1 | 1 | 2
  Other (Medicaid and Medicare) | 0 | 1 | 1
  No insurance | 1 | 0 | 1
Born in the United States [Count of Participants; unit: Participants] | 18 | 21 | 39
Years lived in the United States [Mean (Standard Deviation); unit: Years] | 39.84 (11.6) | 45.38 (12.5) | 42.75 (12.3)
Health comorbidity [Count of Participants; unit: Participants]
  Depression | 6 | 5 | 11
  Psychoses ( | 0 | 4 | 4
  Drug use | 0 | 0 | 0
  Alcohol use | 0 | 1 | 1
  Heart conditions | 0 | 1 | 1
  Diabetes | 6 | 6 | 12
  Hypertension | 2 | 2 | 4
  Cancer | 0 | 0 | 0
  Neurological disorders | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PCL-5 Symptom Score
Description: total count of 20 PTSD symptom ratings on the 0-4 PTSD Checklist for DSM-5 (PCL-5), range = 0=80, higher scores mean a worse outcome
Time Frame: 0 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
Number analyzed (Participants) | 19 | 21
score on a scale | 73.32 (13.7) | 72.95 (14.3)

2. Primary Outcome: Provisional PTSD Diagnosis
Description: count/percent of patients with a provisional diagnosis of PTSD (exceeded a cutoff of 32 and endorsed the required symptoms in each cluster as "Moderately" or higher in frequency following the DSM-5 diagnostic rule)
Time Frame: 0 months
Measure: Count of Participants; unit: Participants
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
Number analyzed (Participants) | 19 | 21
Participants | 19 | 21

3. Primary Outcome: PCL-5 Symptom Score
Description: total count of PTSD symptom scores on the 0-4 PTSD Checklist for DSM-5 (PCL-5), range = 0=80, higher scores mean a worse outcome
Time Frame: approximately 9 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
Number analyzed (Participants) | 19 | 21
score on a scale | 37.07 (17.8) | 47.27 (15.5)

4. Primary Outcome: Provisional PTSD Diagnosis
Description: as for outcome 2
Time Frame: approximately 9 months
Measure: Count of Participants; unit: Participants
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
Number analyzed (Participants) | 19 | 21
Participants | 8 | 14

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | PTSD Care Management (PCM) | Minimally Enhanced Usual Care (MEU)
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/19 | 5/21
Other Adverse Events (participants affected / at risk) | 1/19 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTSD Care Management (PCM) (N=19) | Minimally Enhanced Usual Care (MEU) (N=21)
Severe or significant emotional or psychological distress (Psychiatric disorders) | 3 (3) | 5 (5)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTSD Care Management (PCM) (N=19) | Minimally Enhanced Usual Care (MEU) (N=21)
Release of PII (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
This pilot study was limited to a single clinic and may only generalize to settings that serve African Americans in New Orleans. The small sample size limits statistical conclusion validity, but patients were randomized to each arm so that internal validity was retained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-09-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT03591107/Prot_SAP_000.pdf
  • Informed Consent Form (2018-09-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT03591107/ICF_001.pdf